CLINICAL TRIAL: NCT03776825
Title: Use of Permacol Paste in Perianal Crohn's Disease
Brief Title: Permacol Paste in Perianal Crohn's Disease
Acronym: UPpCro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 2134
Record Dates: First submitted 2018-06-08; First posted 2018-12-17 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Crohn Disease; Perianal Fistula
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Perianal Crohn's Disease: Permacol Paste injection
  Interventions: Device: Permacol Paste

INTERVENTIONS:
Device: Permacol Paste — Permacol Paste Injection

SUMMARY:
The purpose of this study is to collect data about the efficacy of Permacol Paste treatment in perianal Crohn's Disease.

DETAILED DESCRIPTION:
This is an observational prospective cohort study aimed to assess the efficacy of Permacol Paste treatment in perianal Crohn's Disease, by evaluating the healing rate and quality of life of 20 patients prospectively indicated to Permacol Paste treatment during one year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, any sex
* Diagnosis of CD at least 6 months earlier in accordance with clinical, endoscopic, histological an/or radiological criteria
* Presence of perianal fistulas with maximum 3 external openings and a maximum of 2 internal openings, assessed by physical examination and MRI
* Non-active or mildly active luminal CD defined by a CDAI < 220

Exclusion Criteria:

* CDAI > 220
* Dominant luminal active CD requiring immediate surgical or medical therapy
* Fistula with > 3 external openings and > 2 internal openings
* Severe active proctitis and/or rectal stenosis
* Abscess or pelvic collection > 2 cm diameter
* Concomitant rectovaginal fistulas
* Concomitant steroid treatment or treated with steroids in the last 4 weeks

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Perianal Crohn's Disease Patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Perianal fistula closure rate | 12 months
  Complete fistula closure will be defined as absence of spontaneous suppuration or suppuration on applying gentle pressure

SECONDARY OUTCOMES:
Patients quality of life | 12 months
  Quality of life will be assessed using the Inflammatory Bowel Disease Quality of Life (IBDQ). IBDQ is a disease-specific questionnaire included 32 questions. The questions consisted of 4 domains as follows: Bowel symptoms (10 questions), systemic symptoms (5 questions), emotional functioning (12 questions), and social functioning (5 questions). Every question score ranged from 1 to 7 which 7 corresponded to the highest level of functioning. Total score ranged from 32 to 224. Higher score showed higher quality of life.
Patients continence | 12 months
  Continence will be assessed by means of the Cleveland Clinic Incontinence Score (CCIS, or Wexner scale). This scoring system cross-tabulates frequencies and different anal incontinence presentations (Gas/Liquid/Solid/Pad use/Need for lifestyle alterations) and sums the returned score to a total of 0-20 (where 0 = perfect continence and 20 = complete incontinence).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] La Raja C, Maroli A, Foppa C, Gabbiadini R, Dal Buono A, Armuzzi A, Carvello M, Spinelli A. Collagen Paste Injection in Crohn's Disease Perianal Fistula: Long-term Outcomes of a Pilot, Prospective Cohort Study. J Anus Rectum Colon. 2024 Oct 25;8(4):271-278. doi: 10.23922/jarc.2024-008. eCollection 2024. PMID 39473704